CLINICAL TRIAL: NCT00820352
Title: Endothelin Receptor Blockade in Heart Failure With Diastolic Dysfunction and Pulmonary Hypertension
Brief Title: Safety and Efficacy of Bosentan in Patients With Diastolic Heart Failure and Secondary Pulmonary Hypertension
Acronym: BADDHY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Teaching Hospital Hall in Tirol (Other)
Responsible Party: Principal Investigator, Wilhelm Grander, M.D., principal investigator, University Teaching Hospital Hall in Tirol
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BO-001; EUDRACT Number: 2008-005514-40
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Heart Failure, Diastolic; Hypertension, Pulmonary
Keywords: HFNEF; HFPEF; Secondary Pulmonary Hypertension; Endothelin Receptor Blockade
MeSH Terms: conditions — Heart Failure, Diastolic; Hypertension, Pulmonary | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bosentan (Active Comparator): Patients in this arm receive bosentan twice a day for 12 weeks
  Interventions: Drug: bosentan
- placebo (Placebo Comparator): patients in this arm receive 12 placebo twice a day for 12 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bosentan — 4 weeks of oral bosentan 62,5 mg b.i.d., followed by 8 weeks of 125 mg b.i.d.
  Other Names: Ro 47.0203
  Arms: bosentan
Drug: placebo — placebo twice a day for 12 weeks
  Arms: placebo

SUMMARY:
Heart failure is a major medical and socioeconomic problem in western industrial countries, especially with aging populations. Heart failure with normal left ventricle systolic function (heart failure with preserved ejection fraction, HFPEF, heart failure with normal ejection fraction, HFNEF) are common causes of hospitalization mainly in the elderly population and are frequently associated with pulmonary hypertension. It is commonly seen, that patients with left heart disease and pulmonary hypertension with right ventricle dysfunction have a worse prognosis.

The investigators hypothesize, that an additional treatment with Bosentan in this patients will improve their exercise capacity, symptoms, hemodynamics and quality of life.

DETAILED DESCRIPTION:
Heart Failure with preserved ejection fraction is with more than 50% of cases the most common form of heart failure. Typically patients are elderly women with arterial hypertension. Mortality, hospitalization rates due to heart failure and in-hospital complications do not differ significantly from patients with systolic heart failure. However there are some subgroups of HFPEF-patients with a worse prognosis, for example up to 30% of patients develop secondary pulmonary hypertension and thus right ventricle dysfunction. Increased right-ventricle systolic pressure is associated with increased mortality in patients with all forms of heart failure.

There is a lack of evidence about HFPEF. Drugs for treating systolic heart failure showed no improvement in mortality and prognosis. Diuretics are just able to relieve symptoms. There are no clinical trials concerning HFPEF with secondary pulmonary hypertension.

The endothelin system is not only activated in PAH, but also in pulmonary venous hypertension and congestive heart failure, where ET-1 levels rise with the severity of secondary pulmonary hypertension. Pulmonary congestion leads to endothelial dysfunction that results in increased levels of Endothelin-1 (ET-1).

ET-1 is a potent vasoconstrictor. In pulmonary arterial vessels the ETA receptor is the predominant receptor (ratio of ETA to ET B = 9:1), which is responsible for vasoconstriction and remodeling of the pulmonal vasculature. In heart failure the ETA receptor is upregulated. Elevated plasma ET-1 levels correlate with pulmonary artery pressure (PAP), pulmonary vascular resistance (PVR) and inversely with peak exercise capacity.

Recent clinical and laboratory findings indicate comparable pathophysiological mechanisms in pulmonary hypertension secondary to left ventricular dysfunction and pulmonary arterial hypertension. Yet, despite an expanding application in pulmonary artery hypertension, according to current opinion, the oral dual endothelin (ETA/ETB) antagonist bosentan is not indicated for PVH caused by left ventricle / left atrial pressure overload and preserved systolic function. However, there are several studies which show some effects of pulmonary vessel dilating drugs in PAH and left ventricle dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Clinically signs or history of congestive heart failure NYHA II-III (Fatigue, dyspnea on exertion, lung crepitations, pulmonary edema, ankle and or lower leg swelling, jugular pressure enhancement, hepatomegaly)
* Echocardiographic signs of diastolic dysfunction (heart failure with normal ejection fraction)
* Right ventricle enlargement with pulmonary hypertension
* 6 minute walking distance > 150 m < 400 m
* Right Heart Catheterization: Mean PAP > 25 mmHg, PCWP > 15 mmHg

Echocardiographic requirements for definition of heart failure with normal ejection fraction

* E/E' > 15, or
* E/E' > 8 + NTpBNP > 220 pg/ml, or
* E/E' > 8 + E:A < 0.5 + DT > 280 ms or
* Ard-Ad > 30 ms or
* atrial enlargement or
* atrial fibrillation
* NTpBNP > 220 pg/ml + combination
* IVRT - IVRTm < 0 septal und lateral

Echocardiographic requirements for pulmonary hypertension and right ventricle dysfunction

* RVEDD > 30 mm short axis parasternal, and
* one of the following:

  * Tricuspid valve regurgitation velocity (TRV) > 3 m/s;
  * RV-annular systolic velocity < 10 cm/sec (TDI)
  * TAPSE < 18 mm

Exclusion Criteria:

* Patients who are not on guideline conform treatments for cardiovascular disease.
* Left ventricle systolic dysfunction (EF < 50 %), aortic stenosis with peak gradient (instantane) > 40 mm Hg,moderate and severe aortic insufficiency
* moderate and severe mitral regurgitation,
* acute coronary disease, stable coronary artery disease or peripheral vascular disease limiting exercise.
* Other causes of pulmonary - artery - hypertension:

  * relevant obstructive ventilatory disease > grade II (lung functions tests)
  * collagen disease (Tests: MSCT and ANA, ANCA),
  * chronic thrombo- embolic pulmonary arterial hypertension (MSCT),
  * sleep disorder.
  * HIV, HCV, HBV infection.
  * Drug related PAH.
* Orthopaedic disease, immobility, inability to perform 6MWT and cancer.
* Liver disease Child-Pugh B and C, three fold above normal elevated liver enzymes,
* anaemia Hb < 10 mg/dl,
* other specific treatment of pulmonary arterial hypertension including other endothelin receptor blockers, phosphodiesterase inhibitors, prostaglandins and L-arginin
* drug therapy with glibenclamide, rifampicin, tacrolimus, sirolimus, cyclosporine A
* known adverse reactions to bosentan and
* pregnancy and lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
change in 6 minute waling distance after 12 weeks of bosentan (or placebo) treatment | 12 weeks

SECONDARY OUTCOMES:
change in 6 minute walking distance after 24 weeks (12 weeks bosentan or placebo treatment and 12 weeks follow-up) | 24 weeks
changes in hemodynamics assessed by echocardiography after 12 and 24 weeks | 24 weeks
time to clinical worsening after 12 and 24 weeks | 24 weeks
levels of NTpBNP, CRP and Endothelin-1 after 12 and 24 weeks | 24 weeks
Quality of Life assessment (SF-36 and Minnesota Living With Heart Failure Score) after 12 and 24 weeks | 24 weeks
Adverse event count after 12 and 24 weeks | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Grander, M.D., Principal Investigator — University Teaching Hospital Hall i.T.
Locations (7):
- Austria (7):
  - Hospital Mostviertel Waidhofen/Ybbs, Waidhofen an der Thaya, Lower Austria
  - University Teaching Hospital Hall i.T., Hall I. T., Tyrol
  - University Teaching Hospital of the Elisabethinen, Linz, Linz, Upper Austria
  - Hospital Wels/Grieskirchen, Wels, Upper Austria
  - Hospital Hohenems, Hohenems
  - Hospital Natters, Natters
  - University Hospital Salzburg, Salzburg

REFERENCES:
- [Background] Kjaergaard J, Akkan D, Iversen KK, Kjoller E, Kober L, Torp-Pedersen C, Hassager C. Prognostic importance of pulmonary hypertension in patients with heart failure. Am J Cardiol. 2007 Apr 15;99(8):1146-50. doi: 10.1016/j.amjcard.2006.11.052. Epub 2007 Mar 8. PMID 17437745
- [Background] Owan TE, Hodge DO, Herges RM, Jacobsen SJ, Roger VL, Redfield MM. Trends in prevalence and outcome of heart failure with preserved ejection fraction. N Engl J Med. 2006 Jul 20;355(3):251-9. doi: 10.1056/NEJMoa052256. PMID 16855265
- [Background] Shah SJ, Gheorghiade M. Heart failure with preserved ejection fraction: treat now by treating comorbidities. JAMA. 2008 Jul 23;300(4):431-3. doi: 10.1001/jama.300.4.431. No abstract available. PMID 18647986
- [Background] Sanderson JE. Heart failure with a normal ejection fraction. Heart. 2007 Feb;93(2):155-8. doi: 10.1136/hrt.2005.074187. Epub 2005 Dec 30. PMID 16387829
- [Background] Yip GW, Wang M, Wang T, Chan S, Fung JW, Yeung L, Yip T, Lau ST, Lau CP, Tang MO, Yu CM, Sanderson JE. The Hong Kong diastolic heart failure study: a randomised controlled trial of diuretics, irbesartan and ramipril on quality of life, exercise capacity, left ventricular global and regional function in heart failure with a normal ejection fraction. Heart. 2008 May;94(5):573-80. doi: 10.1136/hrt.2007.117978. Epub 2008 Jan 20. PMID 18208835
- [Background] Bhatia RS, Tu JV, Lee DS, Austin PC, Fang J, Haouzi A, Gong Y, Liu PP. Outcome of heart failure with preserved ejection fraction in a population-based study. N Engl J Med. 2006 Jul 20;355(3):260-9. doi: 10.1056/NEJMoa051530. PMID 16855266
- [Background] Bursi F, Weston SA, Redfield MM, Jacobsen SJ, Pakhomov S, Nkomo VT, Meverden RA, Roger VL. Systolic and diastolic heart failure in the community. JAMA. 2006 Nov 8;296(18):2209-16. doi: 10.1001/jama.296.18.2209. PMID 17090767
- [Background] Tribouilloy C, Rusinaru D, Mahjoub H, Souliere V, Levy F, Peltier M, Slama M, Massy Z. Prognosis of heart failure with preserved ejection fraction: a 5 year prospective population-based study. Eur Heart J. 2008 Feb;29(3):339-47. doi: 10.1093/eurheartj/ehm554. Epub 2007 Dec 22. PMID 18156618
- [Background] Sweitzer NK, Lopatin M, Yancy CW, Mills RM, Stevenson LW. Comparison of clinical features and outcomes of patients hospitalized with heart failure and normal ejection fraction (> or =55%) versus those with mildly reduced (40% to 55%) and moderately to severely reduced (<40%) fractions. Am J Cardiol. 2008 Apr 15;101(8):1151-6. doi: 10.1016/j.amjcard.2007.12.014. Epub 2008 Feb 20. PMID 18394450
- [Background] Onishi K, Ohno M, Little WC, Cheng CP. Endogenous endothelin-1 depresses left ventricular systolic and diastolic performance in congestive heart failure. J Pharmacol Exp Ther. 1999 Mar;288(3):1214-22. PMID 10027861
- [Background] Moraes DL, Colucci WS, Givertz MM. Secondary pulmonary hypertension in chronic heart failure: the role of the endothelium in pathophysiology and management. Circulation. 2000 Oct 3;102(14):1718-23. doi: 10.1161/01.cir.102.14.1718. PMID 11015353
- [Background] Lewis GD, Shah R, Shahzad K, Camuso JM, Pappagianopoulos PP, Hung J, Tawakol A, Gerszten RE, Systrom DM, Bloch KD, Semigran MJ. Sildenafil improves exercise capacity and quality of life in patients with systolic heart failure and secondary pulmonary hypertension. Circulation. 2007 Oct 2;116(14):1555-62. doi: 10.1161/CIRCULATIONAHA.107.716373. Epub 2007 Sep 4. PMID 17785618
- [Background] Galie N, Manes A, Branzi A. The endothelin system in pulmonary arterial hypertension. Cardiovasc Res. 2004 Feb 1;61(2):227-37. doi: 10.1016/j.cardiores.2003.11.026. PMID 14736539
- [Background] Cowburn PJ, Cleland JG. Endothelin antagonists for chronic heart failure: do they have a role? Eur Heart J. 2001 Oct;22(19):1772-84. doi: 10.1053/euhj.2000.2557. No abstract available. PMID 11549299
- [Background] Cowburn PJ, Cleland JG, McDonagh TA, McArthur JD, Dargie HJ, Morton JJ. Comparison of selective ET(A) and ET(B) receptor antagonists in patients with chronic heart failure. Eur J Heart Fail. 2005 Jan;7(1):37-42. doi: 10.1016/j.ejheart.2004.08.001. PMID 15642529
- [Background] Opitz CF, Ewert R, Kirch W, Pittrow D. Inhibition of endothelin receptors in the treatment of pulmonary arterial hypertension: does selectivity matter? Eur Heart J. 2008 Aug;29(16):1936-48. doi: 10.1093/eurheartj/ehn234. Epub 2008 Jun 17. PMID 18562303
- [Background] Galie N, Beghetti M, Gatzoulis MA, Granton J, Berger RM, Lauer A, Chiossi E, Landzberg M; Bosentan Randomized Trial of Endothelin Antagonist Therapy-5 (BREATHE-5) Investigators. Bosentan therapy in patients with Eisenmenger syndrome: a multicenter, double-blind, randomized, placebo-controlled study. Circulation. 2006 Jul 4;114(1):48-54. doi: 10.1161/CIRCULATIONAHA.106.630715. Epub 2006 Jun 26. PMID 16801459
- [Background] Rubin LJ, Badesch DB, Barst RJ, Galie N, Black CM, Keogh A, Pulido T, Frost A, Roux S, Leconte I, Landzberg M, Simonneau G. Bosentan therapy for pulmonary arterial hypertension. N Engl J Med. 2002 Mar 21;346(12):896-903. doi: 10.1056/NEJMoa012212. PMID 11907289
- [Background] Sitbon O, Badesch DB, Channick RN, Frost A, Robbins IM, Simonneau G, Tapson VF, Rubin LJ. Effects of the dual endothelin receptor antagonist bosentan in patients with pulmonary arterial hypertension: a 1-year follow-up study. Chest. 2003 Jul;124(1):247-54. doi: 10.1378/chest.124.1.247. PMID 12853530
- [Background] Zolk O, Quattek J, Sitzler G, Schrader T, Nickenig G, Schnabel P, Shimada K, Takahashi M, Bohm M. Expression of endothelin-1, endothelin-converting enzyme, and endothelin receptors in chronic heart failure. Circulation. 1999 Apr 27;99(16):2118-23. doi: 10.1161/01.cir.99.16.2118. PMID 10217651